CLINICAL TRIAL: NCT02119520
Title: PLATELET RICH FIBRIN COMBINED WITH 1.2% ATORVASTATIN FOR TREATMENT OF INTRABONY DEFECTS IN CHRONIC PERIODONTITIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2011-2012/D
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Periodontitis
Keywords: Periodontitis; Surgery; Growth Factors; Statins
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Platelet rich fibrin + atorvastatin (Active Comparator): In Platelet rich fibrin+ATV group PRF combined with 10 µl of 1.2% ATV was inserted into the depth of the IBD
  Interventions: Drug: Platelet rich fibrin +Atorvastatin
- Platelet rich fibrin (Sham Comparator): In Platelet rich fibrin group PRF was inserted into the depth of the IBD.
  Interventions: Drug: Platelet rich fibrin
- Open flap debridement (Other): open flap debridement was followed by no grafting or regenerative intervention.
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Drug: Platelet rich fibrin +Atorvastatin
  Arms: Platelet rich fibrin + atorvastatin
Drug: Platelet rich fibrin
  Arms: Platelet rich fibrin
Procedure: open flap debridement
  Arms: Open flap debridement

SUMMARY:
Current study was designed to evaluate the combined efficacy of PRF and 1.2% ATV gel with open flap debridement (OFD) in treatment of intrabony defects in chronic periodontitis subjects.

ELIGIBILITY:
Inclusion Criteria:

the presence of 3- wall IBD ≥3 mm deep (distance between alveolar crest and base of the defect on an intraoral periapical radiograph [IOPA]) along with an interproximal probing depth (PD) ≥5 mm after phase I therapy (scaling and root planing [SRP]) in asymptomatic teeth.

Exclusion Criteria:

1) Agressive Periodontitis subjects; 2) Systemic conditions known to affect the periodontal status; 3) medications known to affect the outcomes of periodontal therapy; 4) Hematological disorders and insufficient platelet count (<200,000/mm3); 5) pregnancy/lactation; and 6) Smoking and tobacco use in any form 7) Immunocompromised individuals.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage radiographic defect depth reduction | 9 months from baseline
  Defect depth reduction will be assessed from baseline to 9 month post operatively on radiographs

SECONDARY OUTCOMES:
change in probing depth | 9 months from baseline
  probing depth will be assessed from gingival margin to pocket depth at baseline and 9 months postoperatively
change in relative attachment level | 9 months from baseline
  RAL will be assesed from fixed point on the stent at baseline and 9 months postoperatively
change in plaque levels | 9 months from baseline
  plaque levels were assessed at baseline and 9 months postoperatively
change in gingival bleeding | 9 months from baseline
  gingival bleeding was assesed at baseline and 9 months postoperatively
change in gingival margin levels | 9 months from baseline
  change in gingival margin levels were assesed at baseline and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Avani R Pradeep, MDS, Principal Investigator — Professor
Locations (1):
- Govt dental college and research institute, Bangalore, Karnataka, India